CLINICAL TRIAL: NCT05537038
Title: A Phase Ia, Randomized, Placebo-controlled, Double-blind, Dose-finding Evaluation Trial to Describe the Safety, Reactogenicity, and Immunogenicity of Two Investigational Vaccines Against Tuberculosis in IGRA-negative, BCG naïve Subjects
Brief Title: Safety and Immune Responses After Vaccination With Two Investigational RNA-based Vaccines Against Tuberculosis in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: BioNTech SE (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Prevention
Other Study IDs: BNT164-01; 2022-000911-29 (EudraCT Number); 2023-509515-89-00 (EU CTIS Number)
Record Dates: First submitted 2022-09-08; First posted 2022-09-13 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Tuberculosis
Keywords: Prevention of active tuberculosis; RNA Vaccine; Vaccine
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blinded trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- BNT164a1 (Experimental): Escalating dose levels
  Interventions: Biological: BNT164a1
- BNT164b1 (Experimental): Escalating dose levels
  Interventions: Biological: BNT164b1
- Placebo (Experimental): Isotonic NaCl solution (0.9%)
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: BNT164a1 — Multi-antigen ribonucleic acid (RNA) vaccine for active immunization against tuberculosis administered as intramuscular injection
  Arms: BNT164a1
Biological: BNT164b1 — Multi-antigen ribonucleic acid (RNA) vaccine for active immunization against tuberculosis administered as intramuscular injection
  Arms: BNT164b1
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This randomized, placebo-controlled, double-blind, safety and dose-finding Phase Ia trial will evaluate four dose levels of the BNT164 investigational vaccines (BNT164a1 and BNT164b1) to select a safe and tolerable dose in a three-dose schedule.

DETAILED DESCRIPTION:
Enrollment for BNT164a1 and BNT164b1 will be conducted independently, and in parallel. The trial will enroll participants divided into eight dose groups by dose level (4 dose levels per vaccine, i.e., BNT164a1 and BNT164b1) who will be randomized 7:1 to BNT164 (BNT164a1 or BNT164b1):placebo. The trial will use a staggered dose escalation schema with sentinel participants for Dose 1 in all dose groups. The first dose escalation decision will be made based on data from the first 8 participants. The second dose escalation decision will take into account all safety data from participants enrolled in that group. All safety data, e.g., from the 16 participants in the first dose level, will be used for making decisions at higher dose levels.

ELIGIBILITY:
Inclusion Criteria:

* Have given informed consent by signing and dating an informed consent form (ICF) before initiation of any trial-specific procedures.
* Are 18 to 55 years of age inclusive and have a body mass index (BMI) over 18.5 kg/m^2 and under 35 kg/m^2 and weigh at least 50 kg.
* Are willing and able to comply with scheduled visits, treatment schedule, laboratory tests, lifestyle restrictions, and other requirements of the trial. This includes that they are able to understand and follow trial-related instructions.
* Are overall healthy in the clinical judgment of the investigator based on the medical history, clinical assessment (including physical examination, vital signs, clinical laboratory tests, and 12-lead electrocardiogram [ECG]), and be interferon gamma release assay (IGRA)-negative for tuberculosis.
* Hemoglobin ≥12.0 g/dL for volunteers who were born female, ≥13.0 g/dL for volunteers who were born male.
* Volunteers of childbearing potential (VOCBP) that have a negative serum beta-human chorionic gonadotropin pregnancy test result at Visit 0 and negative urine pregnancy test results before each Investigational medicinal product (IMP) injection. Volunteers born female that are postmenopausal (confirmed by follicle stimulating hormone [FSH]) or permanently sterilized (verified by medical records) will not be considered VOCBP.
* VOCBP who agree to practice a highly effective form of contraception and to require their male partners to use condoms, starting at Visit 0 and continuously until 90 days after receiving their last IMP injection in this trial.
* VOCBP who agree not to donate eggs (ova, oocytes) for the purposes of assisted reproduction during trial, starting at Visit 0 and continuously until 90 days after receiving their last IMP injection in this trial.
* Men who are sexually active with a partner of childbearing potential and have not had a vasectomy who agree to use condoms and to practice a highly effective form of contraception during the trial, starting at Visit 0 and continuously until 90 days after receiving their last IMP injection in this trial.
* Men who are willing to refrain from sperm donation, starting at Visit 0 and continuously until 90 days after receiving their last IMP injection in this trial.
* Negative alcohol breath test at Visit 0 or Visit 1.
* With no current use and no history of drug abuse (for amphetamines, benzodiazepines, barbiturates, cocaine, cannabinoids, opiates, methadone, methamphetamines, phencyclidine, tricyclic antidepressants) that in the opinion of the investigator may jeopardize participants' participation and integrity of the trial results.

Exclusion Criteria:

* Any existing condition which may affect vaccine injection and/or assessment of local reactions assessment at the injection site, e.g., tattoos, severe scars, etc.
* Any bleeding diathesis or condition associated with prolonged bleeding that would, in the opinion of the investigator, contraindicate intramuscular injection.
* History of prior tuberculosis vaccination (Bacillus Calmette-Guérin), Mycobacterium tuberculosis infection, treatment for tuberculosis, or history of mycobacterial disease including non-tuberculous mycobacterial infections.
* Current febrile illness (body temperature ≥38.0°C) or other acute illness within 48 hours prior to Dose 1 in this trial (if presented at Visit 0, temporary deferral is allowed).
* History of cardiovascular diseases (diagnosed within the last 3 years), e.g., myocardial infarction, congestive heart failure, cardiomyopathy, clinically significant arrhythmias, myocarditis, or pericarditis.
* History of syncope (fainting) in association with administration of injectable vaccines.
* Known or suspected immunodeficiency.
* History of severe adverse reaction associated with a vaccine and/or severe allergic reaction (e.g., anaphylaxis) to any component of the trial IMP.
* Positive test result at Visit 0 or history of hepatitis B, hepatitis C, or human immunodeficiency virus (HIV).
* Any planned non-trial vaccinations within 28 days before Dose 1 and continuously until 28 days after Dose 3 (Visit 9).

  * Note: Licensed vaccines (including inactivated, mRNA, and live attenuated vaccines) are allowed to be given at least 28 days before or 28 days after each IMP injection.
* Current or planned treatment with immunosuppressive therapy, including systemic corticosteroids (if systemic corticosteroids are administered for ≥14 days at a dose of ≥20 mg/day of prednisone or equivalent) starting at Visit 0 and continuously until 28 days after Dose 3 (Visit 9), for an autoimmune disease. Intraarticular, intrabursal, or topical (skin or eyes) corticosteroids are permitted.
* Have received or plan to receive blood/plasma products or immunoglobulin from 120 days before Dose 1 and continuously until 28 days after Dose 3 (Visit 9).
* Use of any non-trial IMP within 28 days before Dose 1 (Visit 1) in this trial or planned receipt continuously until Visit 12 in this trial, or participation in the active treatment phase of another interventional clinical trial.
* Are subject to exclusion periods from another investigational clinical trial.
* Are breastfeeding or are planning pregnancy or to father children during the trial or within 90 days after Dose 3 in this trial.
* Any screening hematology and/or blood chemistry laboratory value that meets the definition of a Grade >1 abnormality at Visit 0.

  * Note: Trial participants with Grade ≤1 abnormalities (according to the toxicity grading scale) may be considered eligible at the discretion of the investigator.
* Any medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality that, in the investigator's judgment, make the participant inappropriate for the trial.
* Have a history of alcohol abuse or drug addiction within 1 year before Visit 0, or have a history (within the past 5 years) of substance abuse which in the opinion of the investigator, could compromise their wellbeing if they participate as participants in the trial, or that could prevent, limit, or confound the protocol specified assessments.
* Are vulnerable individuals as per International Council on Harmonisation (ICH) E6 definition, i.e., are individuals whose willingness to volunteer in a clinical trial may be unduly influenced by the expectation, whether justified or not, of benefits associated with participation, or of a retaliatory response from senior members of a hierarchy in case of refusal to participate.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2023-04-18 (Actual); Primary Completion 2025-06-06 (Actual); Study Completion 2025-12-08 (Actual)

PRIMARY OUTCOMES:
Frequency of solicited local reactions (pain, erythema/redness, induration/swelling) at the injection site up to 7 days after each dose | Up to 7 days after each dose
Frequency of solicited systemic reactions (vomiting, diarrhea, headache, fatigue, muscle pain and joint pain, chills, and fever) up to 7 days after each dose | Up to 7 days after each dose
Proportion of participants with at least one adverse event (AE) occurring from each dose to 28 days after each dose | From Day 1 until Day 197
Proportion of participants with at least one AE occurring from Dose 1 to 28 days post-Dose 3 | From Day 1 until Day 197
Proportion of participants with at least one serious adverse event (SAE) or medically attended adverse event (MAAE) occurring from Dose 1 up to 168 days post-Dose 3 | From Day 1 until Day 337
Number of AEs from Dose 1 to 28 days post-Dose 3 | From Day 1 until Day 197

CONTACTS AND LOCATIONS:
Overall Officials: BioNTech Responsible Person, Study Director — BioNTech SE
Locations (3):
- Germany (3):
  - emovis GmbH, Berlin
  - CRS Clinical Research Services Berlin GmbH, Berlin
  - CRS Clinical Research Services Mannheim GmbH, Mannheim

IPD SHARING:
Plan to Share IPD: No